CLINICAL TRIAL: NCT03006159
Title: A Phase 1, Randomized, Placebo-controlled, Multiple Dose Escalation Study to Investigate Safety, Pharmacokinetics, and Pharmacodynamics of SHR0534 in Chinese Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0534-Ib
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetic Patients
MeSH Terms: interventions — SHR0534

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Twelve Type 2 Diabetic Patients were randomized in 5:1 ratio to receive multiple (30 days) oral dose of 5 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 2 (Experimental): Twelve Type 2 Diabetic Patients were randomized in 5:1 ratio to receive multiple (30 days) oral dose of 10 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 3 (Experimental): Twelve Type 2 Diabetic Patients were randomized in 5:1 ratio to receive multiple (30 days) oral dose of 25 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo

INTERVENTIONS:
Drug: SHR0534
Drug: Placebo

SUMMARY:
This is a randomized, placebo-controlled, multiple dose escalation study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR0534. The study will be conducted with dose of 5 mg, 10mg and 25 mg. Chinese Type 2 Diabetic patients will be randomized in each cohort to receive the study drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed for more than 3 months;
* HbA1c between ≥7.0 and ≤10.5% for naive patients, or ≥6.5 and ≤9.5% for patients treated with single oral drug, with FPG ≤13.9 mmol/L at randomization;
* Body Mass Index (BMI) between 18 and 40 kg/m^2 (inclusive) with a total body weight of at least 50 kg;
* Agree to stop any other drugs for diabetes during washout and study period;
* Serum C peptide concentration ≥0.8ng/mL at randomization.

Exclusion Criteria:

* Participated any drug clinical trials within 3 months or ≥3 times during the last year, or had blood donation/loss≥400mL or as Blood recipient within 3 months before randomization;
* History use of Insulin within 6 months;
* Drug or alcohol abuse within 6 months;
* Use any other hypoglycemic drugs or weight reducing drugs within 3 months, or use any grug or dietary supplements within 1 weeks prior to screening ;
* Underwent surgical procedures within 1 month prior to screening, or planned major surgical procedures during the study period;
* Subject who cannot refrain from smoking, eating and/or drinking containing xanthine/caffeine, or strenuous exercise, or others that affect drug absorption, distribution, metabolism and excretion within 2 days before the study drug administration;
* With active hepatitis;
* Uncontrolled endocrine system diseases (such as hyperthyroidism, hypothyroidism, Cushing syndrome, multiple endocrine neoplasia);
* Uncontrolled hypertension with systolic blood pressure (SBP) > 160mmHg and / or diastolic pressure (DBP) > 100 mmHg after drug treatment;
* History of recurrent severe hypoglycemia;
* With severe chronic gastrointestinal disease (e.g., an active ulcer within 6 months) or treatment that may affect drug absorption (e.g., gastrointestinal surgery);
* With any cancer (other than skin basal cell carcinoma) that has been treated or untreated within the last 5 years;
* History of decompensated heart failure (NYHA grade III and IV), unstable angina, stroke or transient ischemic attack, persistent myocardial infarction, and the clinical significance of arrhythmia (such as frequent contractions), or had coronary artery bypass grafting or percutaneous coronary intervention within 6 months;
* History of acute metabolic complications, or proliferative retinopathy or maculopathy which required acute treatment within 6 months;
* Severe trauma or severe infection that may affect glycemic control within 1 months before screening;
* AST, ALT or TBIL>1.5×UNL, or Cre>1.5 mg/dL(male)/1.4 mg/dL(female), or ACR>300mg/g at screening;
* Positive of hepatitis B surface antigen, hepatitis C antibody, HIV antibody or syphilis antibody;
* With clinical significance abnormal of ECGs, such as II or III degree atrioventricular block (except right bundle branch block), long QT syndrome or QTc>500 MS;
* Subject was not suitable for the study as determined by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | From baseline up to 8 days after last treatment (Day 38)
Area under the plasma concentration curve after the first and last multiple oral dose (AUC) | From time 0 to 24 hours for the first dose, and from time 0 to 192 hours after the last dose
Peak plasma concentration (Cmax) after the first and last multiple oral dose | From time 0 to 24 hours for the first dose, and from time 0 to 192 hours after the last dose
Terminal elimination halflife (t½) for SHR0534 after the last multiple oral dose | From time 0 to 192 hours after the last dose
Changes in the concentrations of blood glucose and insulin after multiple oral dose | From baseline up to 24 hours after last treatment (Day 31)]

IPD SHARING:
Plan to Share IPD: No